CLINICAL TRIAL: NCT04483310
Title: Meditation-Relaxation (MR Therapy) for Sleep Paralysis: A Pilot Study in Patients With Narcolepsy
Brief Title: Meditation-Relaxation (MR Therapy) for Sleep Paralysis.
Acronym: MR_Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18090
Record Dates: First submitted 2020-07-03; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Sleep Paralysis; Narcolepsy Type 1
Keywords: Behavioral Treatment; Sleep Paralysis; Narcolepsy Type 1
MeSH Terms: conditions — Sleep Paralysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MR therapy (Experimental): MR therapy is a psychological treatment for SP, comprised of the following steps applied directly during the attack: Step I: Reappraisal of the meaning of the attack; Step II: psychological and emotional distancing; Step III: inward focused-attention meditation; Step IV: Muscle relaxation.
  Interventions: Behavioral: MR therapy.
- Control intervention (Active Comparator): The control intervention was identical, except participants engaged in deep breathing; entailing slow deep breaths, while repeatedly counting from 1-10. This is an active control (breathing-distraction exercise) rather than a placebo.
  Interventions: Behavioral: breathing-distraction exercise

INTERVENTIONS:
Behavioral: MR therapy. — MR therapy is based on 4 steps applied directly during the attack: Step I: Reappraisal of the meaning of the attack; Step II: psychological and emotional distancing; Step III: inward focused-attention meditation; Step IV: Muscle relaxation.
  Arms: MR therapy
Behavioral: breathing-distraction exercise — The control intervention is based on a breathing exercise, the patients should entail slow deep breaths, while repeatedly counting from 1-10
  Arms: Control intervention

SUMMARY:
The aim of the study is to evaluate, with a small-scale pilot study, the efficacy of Meditation Relaxation therapy for Sleep Paralyses in patients with narcolepsy. The study involves two arms, with intervention with Meditation Relaxation therapy or sham over a period of three months.

ELIGIBILITY:
Inclusion Criteria:

* Narcolepsy (type 1 and 2) based on polysomnography, Multiple Sleep Latency Test [MLST] and CSF hypocretin level testing).
* Patients had to have experienced SP at least four times in the last month.

Exclusion Criteria:

* Psychiatric comorbidity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Paralysis Experiences and Phenomenology Questionnaire (SP-EPQ) | Three months.
  The questionnaire addresses the distress associated with SP.

SECONDARY OUTCOMES:
Daily journal | Three months.
  Each day during the study (12 weeks), participants rated their SP occurrence, perceived duration (sec./min.), fear associated with SP, and disturbance caused by hallucinations (on a ten-point scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL di Bologna, Bologna, Italy